CLINICAL TRIAL: NCT06106243
Title: Oral Health-Related Quality of Life and Retention in Digitally Versus Conventionally Fabricated Flexible Removable Partial Dentures in Maxillary Class III Modification 1 Patients: A Cross-over Randomized Clinical Trial
Brief Title: Evaluation of Digital 3D Printed Temporary Removable Partial Denture.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Medhat Sameh Shehata Abdelaziz, PHD student in prosthodontics department, Cairo University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 7-7-23
Record Dates: First submitted 2023-10-24; First posted 2023-10-30 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Partial-edentulism; Temporary Partial Denture; 3D Printing; Oral Health Related Quality of Life

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The conventional heat pressing temporary flexible maxillary removable partial denture (Active Comparator)
  Interventions: Procedure: The conventional heat pressing temporary flexible maxillary removable partial denture
- 3D-printed and digitally designed temporary flexible maxillary removable partial denture . (Experimental)
  Interventions: Procedure: 3D-printed and digitally designed temporary flexible maxillary removable partial denture

INTERVENTIONS:
Procedure: The conventional heat pressing temporary flexible maxillary removable partial denture — An intraoral scan will be made for each patient's maxillary and mandibular jaws in addition to digital bite registration using (Medit i700; Medit corp.) the resultant data will be exported in the form of a Standard Tessellation Language (STL) file. The denture base and the teeth will be designed using computer-aided design software (Partial Cad, Dental CAD software). Each patient will receive two RDPs, fabricated with two different manufacturing techniques. Based on randomization, the patients will start by receiving either partial denture that is fabricated by conventional heat pressing technique of 3D printed castable resin (Cast V1resin) followed by partial denture that is fabricated by 3D printing of printable resin (Flexo denture base, resin) and teeth (permanent crown,resin) or the other way around. In 3D-printed RDP, the artificial teeth will be attached to the fabricated denture bases using printable denture base resin material
  Arms: The conventional heat pressing temporary flexible maxillary removable partial denture
Procedure: 3D-printed and digitally designed temporary flexible maxillary removable partial denture — 3D-printed and digitally designed temporary flexible maxillary removable partial denture
  Arms: 3D-printed and digitally designed temporary flexible maxillary removable partial denture .

SUMMARY:
This study aims to compare oral health-related quality of life and retention between digitally- fabricated temporary flexible RDPs and conventionally-fabricated temporary flexible RDPs.

ELIGIBILITY:
Inclusion Criteria:

* Maxillary Class III, modification I partially edentulous patients that enables measuring the retention values intraorally without denture rotation.
* Fully dentulous or partially edentulous opposing mandibular arch.
* Patients that require temporary partial dentures for aesthetic reasons or as an interim denture during mouth rehabilitation treatment or after implant placement.
* Age range (30-55 years).
* Cooperative patients that are willing to attend all follow-up periods.
* Patients with healthy attached mucosa of appropriate thickness free from any inflammation.
* Patients with healthy abutments and healthy periodontium and no more than grade I mobility.

Exclusion Criteria:

* Patients with Parkinson's disease
* Patients with xerostomia.
* Patients with a history of allergy to dentures made of resins.
* Patients with pathological changes of residual ridges as recurrent or persistent ulcers, osteomyelitis and infections.
* Patients with large irregular bony exostosis.
* Patients with medical or psychological conditions as physical disability or mental retardation that hinder cooperation in the follow up visits and answering the questionnaires.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Estimated)
Dates: Start 2023-06-02 (Actual); Primary Completion 2024-08-02 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Oral health-related quality of life. | Baseline and 6 months
  Oral health impact profile (OHIP 14) questionnaire will be used to asses the oral health-related quality of life
Retention of a removable partial denture | Baseline and 6 months
  The retention will be measured using Digital Force Gauge attached to the denture polished surface while the patient is in supine position

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dentistry , Cairo university, Giza, Egypt